CLINICAL TRIAL: NCT04009538
Title: The Effect of Re-Rehabilitation in Patients With COPD
Brief Title: Re-Rehabilitation in Chronic Obstrctive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ilknur Naz, Asst. Prof., Izmir Katip Celebi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IzmirKCU1
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Copd; Smoking; Smoking Cessation; Rehabilitation; Tobacco Use
Keywords: copd; smoking; Smoking Cessation; Rehabilitation; Tobacco Use
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking; Smoking Cessation; Tobacco Use | interventions — Rehabilitation; Exercise

STUDY DESIGN:
Intervention Model Description: COPD patient participated first and second rehabilitation program
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COPD patients participated PR program (Experimental): COPD patients participated first and second PR program
  Interventions: Other: Rehabilitation program

INTERVENTIONS:
Other: Rehabilitation program — exercise program twice a week
  Other Names: exercise

SUMMARY:
Patients with COPD who participated in the second rehabilitation program in the Pulmonary Rehabilitation unit will be included in the study. Pulmonary function tests, arterial blood gases, mMRC dyspnea perception, 6-minute walking distance, disease-specific (SGRQ) quality of life and hospital anxiety depression scale values will be compared.

DETAILED DESCRIPTION:
Pulmonary rehabilitation (PR) program in patients with COPD reduces dyspnea perception, increases exercise capacity, improves quality of life, and reduces psychological symptoms. Unfortunately, these gains are not permanent, but disappear within 12-24 months. The aim of this study is to compare the gains of the second PR program with the first program.

Patients with COPD who participated in the second rehabilitation program in the Pulmonary Rehabilitation unit will be included in the study. Pulmonary function tests, arterial blood gases, mMRC dyspnea perception, 6-minute walking distance, disease-specific (SGRQ) quality of life and hospital anxiety depression scale values will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years
* Completed PR program

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Exercise Capacity | 6 minutes
  Six minutes walk test

SECONDARY OUTCOMES:
Respiratory Functions | 30 minutes
  Pulmonary Function Test
Dyspnea Sensation | 5 minutes
  We used "Modified Medical Research Council (MMRC)" dyspnea scale, which consists of 5 items ranging between 1 and 5, to determine the severity of patients' shortness of breath. The score "1" represents the best level, where the score "5" indicates the poorest.
Disease Specific Quality of Life | 20 minutes
  We used St. George's Respiratory Questionnaire (SGRQ) to determine disease-specific quality of life. At this scale, high scores define worsened disease and increased symptoms.
Anxiety and Depression | 20 minutes
  Hospital Anxiety and Depression (HAD) Inventory was used for assessment of anxiety and depression. In this scale; scores of anxiety and depression are calculated separately. The maximum score for both is 21 and high scores correspond to high degree anxiety and depression. Cut-off scores for anxiety and depression were determined as 10/11 and 7/8 respectively.